CLINICAL TRIAL: NCT04940988
Title: Impacts of a Physician-targeted Price Transparency Real Time Prescription Benefits Tool on Medication Out-of-pocket Costs
Brief Title: Impacts of a Physician-targeted Price Transparency Tool on Medication Out-of-pocket Costs
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-RTPB
Record Dates: First submitted 2021-03-18; First posted 2021-06-28 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Prescriptions; Costs and Cost Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- See alert: The intervention group refers to medication orders placed by prescribers when practicing in an outpatient department randomly assigned to receive the intervention, which is implementation of the RTPB tool.
  Interventions: Other: Real-time benefits check
- Do not see alert: The non intervention group refers to medication orders placed by prescribers when practicing in an outpatient department randomly selected to not receive the intervention.

INTERVENTIONS:
Other: Real-time benefits check — Prescribers practicing in outpatient departments assigned to the intervention arm will be shown popup alerts with their patient's insurance benefit design-specific out-of-pocket cost for the drug being ordered as well as out-of-pocket costs for up to 3 lower-cost alternatives if available. Alternatives will only be shown when available and when the patient and his or her benefit design information can be matched by the electronic health record system to accurately query out-of-pocket cost information.
  Other Names: Physician-focused medication price transparency
  Groups: See alert

SUMMARY:
The goal of this study is to evaluate whether presenting patient out-of-pocket cost information to the provider at the time of prescribing leads to orders for medications with lower out-of-pocket costs. The Real-Time Prescription Benefits (RTPB) tool has been implemented to randomly selected providers across NYU Langone Health's outpatient physician practices. The RTPB tool provides physicians with information about patient out-of-pocket (OOP) cost for medications at the point of outpatient prescribing. OOP is inclusive of any copay, coinsurance, and deductible that the patient owes given their prescription drug benefit plan. If the physician is submitting a prescription order and a clinically-appropriate alternative with a lower OOP cost is available, an alert with OOP cost information for the drug being initially ordered as well as up to three lower-cost alternatives will be displayed. Implementation of this tool will be analyzed to see if it will lead to reduced out-of-pocket costs on ordered medications when alternatives were available. Because effects could vary along many dimensions (e.g., specialty, drug class, insurance type), secondary analyses will be conducted and stratified along such dimensions. Analyses will be conducted at the prescription order level.

ELIGIBILITY:
Inclusion Criteria:

* Medication orders for which this match and query was successful and outcomes data was available.

Exclusion Criteria:

* No patient-level exclusion criteria will be imposed

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The intervention group refers to medication orders placed by prescribers when practicing in an outpatient department randomly assigned to receive the intervention, which is implementation of the RTPB tool. The control group refers to medication orders placed by prescribers when practicing in an outpatient department randomly selected to not receive the intervention.
Sampling Method: Probability Sample
Enrollment: 21401 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Medication out of pocket cost per day | Through study completion, an average of 1 year
  The primary outcome, which will be measured at the medication-order level is out-of-pocket cost per day for a drug ordered. It will be computed by dividing the out-of-pocket cost of a drug by the days supply. Data will be collected through the electronic health record.

SECONDARY OUTCOMES:
Whether an order was placed for a mail-order pharmacy | Through study completion, an average of 1 year
  A secondary outcome, also specified at the order level, is whether a drug prescription was ordered from a mail-order pharmacy, since switching to a mail-order pharmacy often presents an opportunity for savings. Data will be collected through the electronic health record.
Days supply | Through study completion, an average of 1 year
  A secondary outcome, also specified at the order level, is the days supply. Data will be collected through the electronic health record.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desai SM, Chen AZ, Wang J, Chung WY, Stadelman J, Mahoney C, Szerencsy A, Anzisi L, Mehrotra A, Horwitz LI. Effects of Real-time Prescription Benefit Recommendations on Patient Out-of-Pocket Costs: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2022 Nov 1;182(11):1129-1137. doi: 10.1001/jamainternmed.2022.3946. PMID 36094537